CLINICAL TRIAL: NCT07138560
Title: BOOST-PD - Better On-time Observations of Motor Fluctuations Using Wearable Sensor Technology: A Naturalistic Study on IPX-203 for Parkinson's Disease
Brief Title: BOOST-PD A Naturalistic Study on IPX-203 for Parkinson's Disease
Acronym: BOOST-PD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Amneal Pharmaceuticals, LLC (Industry)
Responsible Party: Principal Investigator, Hubert Fernandez, Center Director, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-070; 4322795 (Other Grant/Funding Number: Amneal Pharmaceuticals LLC)
Record Dates: First submitted 2025-05-15; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
Keywords: Crexont; motor fluctuations
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Arm (Other): The intervention arm will be patients converting to shorter dose intervals of Crexont (IPX203) and allowing for higher dosing frequency, as practiced in real-world settings, combined with objective monitoring of on-time periods and other parameters using the KinesiaU device, could reveal additional benefits of Crexont (IPX203) treatment.
  Interventions: Drug: CREXONT ER

INTERVENTIONS:
Drug: CREXONT ER — exploring shorter dose intervals of Crexont (IPX203) and allowing for higher dosing frequency, as practiced in real-world settings, combined with objective monitoring of on-time periods
  Other Names: IPX203

SUMMARY:
The purpose of this study is to evaluate the effect of IPX203 (Crexont®) - the newest extended-release levodopa formulation - on the duration and quality of good on time, using a wearable device to monitor symptoms. 'Good on time' refers to a period (minutes to hours) when a patient experiences optimal symptom control due to effective medication and has better overall functioning without troublesome dyskinesias. The change in the duration and quality of on-time will be measured by a wearable device placed on your wrist called KinesiaU.

DETAILED DESCRIPTION:
This research is being done because a new, longer-duration formulation of levodopa named IPX203 (brand name: Crexont®) has been recently approved by the FDA. The pivotal study on this drug demonstrated that IPX203 significantly increased the daily good on-time compared to immediate release carbidopa-levodopa (IR CD-LD), where good on-time is the time when the Parkinson's symptoms are improved without troublesome dyskinesias. In that study, the participants were taking IPX203 a mean of 3 times per day which still left a mean of 4.18 hours of off-time per day (when symptoms returned). These data were based on diaries filled out by the participants.

The aim of the study is to expand the current knowledge on IPX203, analyzing the changes in good on-time after careful and tailored adjustments, as in the real-world setting. This will be done with the assistance of a wearable device to obtain objective data. Additional variables such as changes in the tremor scores, conversion from other drugs such as Rytary and COMT inhibitors, and the difference between starting and final IPX203 doses will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* - Participant is 40 years or older
* Diagnosed with idiopathic Parkinson's disease and is deemed to be levodopa responsive
* Baseline MDS-UPDRS score in OFF-state is > 20
* Patient is being treated with a stable regimen of CD-LD for at least four weeks
* The minimum most frequent levodopa dosing is 100 mg if using IR CD-LD and 195mg if using Rytary; maximum levodopa dosing per day is 1200 mg if using IR CD-LD, 1000 mg if associated with a COMT inhibitor, and 2400 mg if using Rytary
* Participant can be on stable doses of any levodopa adjunctive medications and/or psychotropic medications for at least 30 days
* Participant experiences off time estimated at 2 hours or more per day; participant can comply with the wearable kinematic device.

Exclusion Criteria:

* - Participants with severe dyskinesia as defined by a score of 4 on Question 4.1 (time spent with dyskinesia) of UPDRS IV
* Currently on device-aided therapies for advanced PD
* Using controlled-release CD-LD apart from a single daily bedtime dose
* Using "on demand" therapy unless willing to stop it during the study period
* Have a diagnosis hypothesis of dopamine dysregulation syndrome or evidence of significant levodopa-related complications including orthostatic hypotension or psychosis
* History of dementia or MOCA score lower than 23
* Significant medical history might interfere significantly with study participation
* Being enrolled in other clinical trials involving active medication interventions.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 8 weeks
  Mean change in the average duration of good on-time from baseline to end of study

SECONDARY OUTCOMES:
Secondary Endpoint | 8 weeks
  Mean change in the average 'slowness' scores as measured by KinesiaU
Secondary Endpoint | 8 weeks
  Mean change in time spent with tremor as measured by KinesiaU
Secondary Endpoint | 8 weeks
  Mean change in the average tremor scores as measured by KinesiaU
Secondary Endpoint | 8 weeks
  Mean change in time spent with dyskinesia as measured by KinesiaU
Secondary Endpoint | 8 weeks
  Mean change in the continuous on time as measured by KinesiaU

OTHER OUTCOMES:
Exploratory Endpoints | 8 weeks
  Mean difference between KinesiaU and PD diary measurements of change in good on-time from baseline to end of study
Exploratory Endpoint | 8 weeks
  Difference in the Patient Global Impression of Change from baseline to end of study.
Exploratory Endpoint | 8 weeks
  Difference between Non-Motor Fluctuation Assessment Questionnaire from baseline to end of study.
Exploratory Endpoint | 8 weeks
  The average time (in weeks) taken to reach the final dose.
Exploratory Endpoint | 8 weeks
  The average number of adjustments needed to reach the final dose.

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Fernandez, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Modi NB, Mittur A, Dinh P, Rubens R, Gupta S. Pharmacodynamics, Efficacy, and Safety of IPX203 in Parkinson Disease Patients With Motor Fluctuations. Clin Neuropharmacol. 2019 Sep/Oct;42(5):149-156. doi: 10.1097/WNF.0000000000000354. PMID 31306216
- [Background] Hauser RA, Espay AJ, Ellenbogen AL, Fernandez HH, Isaacson SH, LeWitt PA, Ondo WG, Pahwa R, Schwarz J, Stocchi F, Zeitlin L, Banisadr G, Fisher S, Visser H, D'Souza R. IPX203 vs Immediate-Release Carbidopa-Levodopa for the Treatment of Motor Fluctuations in Parkinson Disease: The RISE-PD Randomized Clinical Trial. JAMA Neurol. 2023 Oct 1;80(10):1062-1069. doi: 10.1001/jamaneurol.2023.2679. PMID 37578800
- [Background] Hauser RA, Fernandez HH, Jimenez-Shahed J, Allard S, Banisadr G, Fisher S, D'Souza R. Duration of "Good On" time per dose: Immediate-release carbidopa-levodopa vs. extended-release carbidopa-levodopa (IPX203, CREXONT(R)). Parkinsonism Relat Disord. 2025 Feb;131:107239. doi: 10.1016/j.parkreldis.2024.107239. Epub 2024 Dec 15. PMID 39733558